CLINICAL TRIAL: NCT06648863
Title: Bahir Dar Child Development Study, Ethiopia
Acronym: BCD
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Addis Continental Institute of Public Health (Other); New York University (Other); Boston Children's Hospital, Boston, MA, USA (Other)
Responsible Party: Principal Investigator, Anne Lee, Director Global Newborn Health, Brigham and Women's Hospital
Other Study IDs: 2022P002539
Record Dates: First submitted 2024-10-08; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Development, Child; Behavior, Social
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- A/6 months: Measures of child development (GSED), nutrition, medical history and anthropometrics, followed by MRI
- B/12 months: Measures of child development (GSED), nutrition, medical history and anthropometrics, followed by MRI
- C/18 months: Measures of child development (GSED), nutrition, medical history and anthropometrics, followed by MRI
- D/24 months: Measures of child development (GSED), nutrition, medical history and anthropometrics, followed by MRI
- E/30 months: Measures of child development (GSED), nutrition, medical history and anthropometrics, followed by MRI
- F/36 months: Measures of child development (GSED), nutrition, medical history and anthropometrics, followed by MRI
- G/48 months: Measures of child neurocognitive development and school readiness, nutrition, medical history, and anthropometrics followed by MRI
- H/60 months: Measures of child neurocognitive development and school readiness, nutrition, medical history, and anthropometrics followed by MRI

SUMMARY:
The goal of this observational study is to learn about typical neurodevelopment in children aged 6 months to 5 years who live in Bahir Dar, Ethiopia. The main aims of the study are:

Aim 1: To characterize typical neurodevelopment as measured by i) brain volume using low-field MRI and ii) scores on behavioral assessments of early child neurodevelopment.

Aim 2: To characterize typical pre-academic school skills in early childhood as measured by tasks of visual processing, reasoning, verbal expression and school readiness.

Aim 3: To identify factors influencing child development in a community in Bahir Dar, Amhara region of Ethiopia, as measured by validated measures of maternal mental health, home environment, and childhood adversity.

Participants will complete one low-field MRI scan at enrollment, have a hemoglobin blood test, and undergo age-appropriate neurodevelopmental assessments and surveys that may include:

* WHO Global Scales for Early Development (GSED) [ages 6 - 36 months]
* Tasks of visual reasoning and verbal expression [ages 48-60 months]
* Executive Functions test using the tablet-based NIH Toolbox [ages 48-60 months]
* School Readiness questionnaire assessing knowledge of literacy, numeracy, early reading, crystallized knowledge, memory, and self-regulation [ages 48-60 months]
* Maternal report of child's motor, cognitive and socioemotional skillsChild Anthropometrics assessment

Additional assessments of the participant's family and environment will include

* Medical History questionnaire
* Family socioeconomic status
* Maternal Mental Health
* Recent Life Events and hardship
* Home Environment and Parenting UNICEF's MICs Family Care Indicators)
* Food security and feeding practices

DETAILED DESCRIPTION:
More than 170 million children worldwide under 5 years of age fail to meet their developmental potential . Reduced or impaired neurodevelopment in early life can impact lifelong patterns of cognitive and behavioral development, beginning with early and pre-academic skills that are vital to academic success, achievement, and predictive of later income, health access, and socioeconomic standing. Improved early neurodevelopment, on the other hand, can spark an intergenerational cascade of improved family and child health outcomes.

Infant and early childhood neurodevelopment can be impacted by a diverse array of environmental factors beginning from the earliest stages of fetal development. Premature birth, low birth weight, poor maternal health, maternal stress, inadequate maternal and infant nutrition, reduced breastfeeding, exposure to disease, environmental neurotoxicants, and environmental adversity can all shape developing brain systems and impact emerging brain cognitive and behavioral functions. However, there is a gap in our understanding of neurodevelopmental patterns in children across LMIC settings where many neurodevelopmentally impactful adversities are magnified. Increased knowledge of risk and protective factors associated with neurodevelopmental characteristics in children can support the identification of the global and regional factors that drive poor neurodevelopmental outcomes in children and help to inform interventions to improve child outcomes

The Bahir Dar Child Development (BCD) study will characterize patterns of neurodevelopment in a community sample of children in Bahir Dar, Amhara, Ethiopia using a cross-sectional design covering children aged 6 - 60 months. Neuroimaging data collected using a low-field portable MRI scanner will be coupled with neurocognitive assessments and a broad assessment of child and family medical history, nutritional status, socioeconomic standing, and other social determinants of health. These data will be harmonized and integrated with similar data collected from other regions and countries to provide a global map of development and identify important targetable factors that will improve neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children living in Bahir Dar town with parents who are willing and able to travel to Felege Hiwot Regional Hospital clinic for study visits
* Healthy child without active clinical symptoms/complaints
* Child within specified age ranges for each cohort/group (+/- 2 months)

Exclusion Criteria:

* Child born with a severe congenital birth defect or hypoxic ischemic encephalopathy (birth asphyxia) per maternal report
* Severe developmental or behavioral disorder per maternal report
* Severe illness/clinical signs or symptoms of illness based on maternal and child report (including vomiting, headache, or seizures)
* Plans to move out of catchment area in less than 1 year

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children will be identified at rural health centers, outpatient vaccination clinics or campaigns, and other health facilities around Bahir Dar, Amhara, Ethiopia.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Total Brain MRI volumes | Collected in all children (ages 6-60 months) at enrollment.
  Total supratentorial brain volume measured from Hyperfine MRI uzing standard processing pipelines for infant MRI progressing. Outcomes will be reported in cm3.

SECONDARY OUTCOMES:
WHO Global Scales for Early Development (GSED) | Collected in children aged 6-36 months at enrollment.
  WHO Global Scales for Early Development (GSED) will be administered in both short from (caregiver report) and long form (observarion). Outcomes will be calculate and reported in standardized scores called the DAZ scores, following guidelines provided in the WHO technical report [https://iris.who.int/bitstream/handle/10665/366272/WHO-MSD-GSEDpackage-v1.0-2023.8-eng.pdf]. For each form, we will calculate a total score and scores for subdomains of cognitive, motor, language, and social-emotional development.
Visual reasoning | Collected in children aged 48-60 months at enrollment.
  Visual reasoning will be assessed using a visual matrix completion task. Scores are calculated as total scores ranging from 0-29.
School readiness | Collected in children aged 48-60 months at enrollment.
  School readiness score are based on direct assessment involving questions that assess constructs such as early literacy, numeracy, verbal expression, and crystalized knowledge. Scores are calculated as a total score ranging from 0-25.
Executive Functioning: cognitive flexibility and attention | Collected in children aged 48-60 months at enrollment.
  The dimensional Change Card Sort (DCCS) task will be administered using the NIH toolbox app on an ipad. DCCS measures cognitive flexibility and attention. Children are shown figures (stimuli) that vary across two dimensions, shape and color. The child is asked to select one of two stimuli that best match a central target stimulus based on one characteristic (shape or color). Children practice matching based on color and shape before the actual trial items. Computer-generated scores reflected accuracy and reaction time metrics (see the NIH Toolbox Manual).
Self-regulation | Collected in children aged 48-60 months at enrollment.
  Observer rated score of self-regulation skills adapted from IDELA and the Preschool Self-Regulation Assessment. The scale as 7 items reported on a 4-point Likert scale (1= almost never; 2=Sometimes, 3=Often, 4=Almost always). A total score is creating summing the 7 items to create a scale ranging from 7-28.
Verbal expression | Collected in children aged 48-60 months at enrollment.
  A verbal expression will be assessed using a task of verbal reasoning where the child is asked to descibe a category that captures two objects or phenomena by completing a sentence like "Green and Yellow are both... ?" to which the correct answer is "colors". A total score will be calculated ranging from 0-20.
Executive Functioing: inhibitory control and attention | Collected in children aged 48-60 months at enrollment.
  The Flanker Task (FT) measures inhibitory control and attention. The FT task will be administered using the NIH Toolbox App on an iPad. Children are presented with a row of fish and/or arrows and have to select a response button that shows the direction of the central stimulus (fish or arrow) by pressing one of two buttons on the screen. Computer generated scores reflected accuracy and reaction time metrics (see the NIH Toolbox Manual).
Executive Functioning: processing speed | Collected in children aged 48-60 months at enrollment.
  The Speed matching (SM) task assesses processing speed. The SM task will be administered using the NIH Toolbox App on an iPad. Children are asked to identify which of four targets (pictures of two-dimensional animal faces) match the target picture at the top of the screen by tapping an image as quickly as possible without making mistakes. The task starts with four practice items with feedback. The trial finished after 90 seconds. Computer-generated scores reflected accuracy and reaction time metrics (see the NIH Toolbox Manual).

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Lee, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Yemane Berhane, MD, PhD, Principal Investigator — Addis Continental Institute of Public Health
Locations (1):
- Health Center, Bahir Dar, Addis, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jensen SKG, Yibeltal K, North K, Workneh F, Teklehaimanot A, Abate BH, Fasil N, Melka TL, Chin TI, Folger LV, Roy Paladhi U, Van Dyk F, Thomason ME, Grant PE, Inder T, Worku A, Berhane Y, Lee AC. Bahir Dar Child Development Cross-Sectional Study, Ethiopia: study protocol. BMJ Paediatr Open. 2025 Apr 2;9(1):e003173. doi: 10.1136/bmjpo-2024-003173. PMID 40180427